CLINICAL TRIAL: NCT03541850
Title: Prospective Study of Stereotactic Body Radiotherapy (SBRT) Following Radical Prostatectomy
Brief Title: Stereotactic Body Radiation Therapy in Treating Patients With Localized Prostate Cancer That Have Undergone Surgery
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Viewray Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-001064; NCI-2017-02032 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-04-09; First posted 2018-05-31 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: PSA Level Greater Than 0.03; PSA Progression; Stage I Prostate Adenocarcinoma AJCC (American Joint Committee on Cancer ) v7; Stage II Prostate Adenocarcinoma AJCC v7; Stage III Prostate Adenocarcinoma AJCC v7
MeSH Terms: interventions — Androgen Antagonists; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (SBRT, ADT) (Experimental): Patients undergo SBRT QOD for 14 days. Patients may also receive ADT comprised of a luteinizing hormone-releasing hormone agonist or a gonadotropin-releasing hormone antagonist, and an oral anti-androgen for 6 months at the discretion of the treating physician.
  Interventions: Drug: Antiandrogen Therapy; Other: Quality-of-Life Assessment; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Antiandrogen Therapy — Receive luteinizing hormone-releasing hormone agonist or gonadotropin-releasing hormone antagonist, and oral anti-androgen
  Other Names: ADT; Androgen Deprivation Therapy; Anti-androgen Therapy; Anti-androgen Treatment; Antiandrogen Treatment; Hormone Deprivation Therapy; Hormone-Deprivation Therapy
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This phase II trial studies how well stereotactic body radiation therapy works in treating patients with prostate cancer that has not spread to other parts of the body and have undergone surgery. Stereotactic body radiation therapy is a specialized radiation therapy that sends x-rays directly to the tumor using smaller doses over several days and may cause less damage to normal tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of postoperative stereotactic body radiation therapy (SBRT) at a dose of 34 grays (Gy) in five fractions, as compared with historical control efficacy rates in patients who received conventionally fractionated postoperative radiotherapy.

II. To determine the toxicity of postoperative SBRT at a dose of 34 Gy in five fractions, both via physician-scored and patient-reported metrics.

SECONDARY OBJECTIVES:

I. To determine the proportion of SBRT fractions for which on-line adaptive radiotherapy is required due to changes in organ-at-risk anatomy, in the subset of patients treated with magnetic resonance imaging (MRI)-guided radiotherapy.

II. To gather biomarkers that may elucidate predictors of increased efficacy or increased toxicity.

TERTIARY OBJECTIVES:

I. To compare toxicity profiles (both physician-scored and patient-reported) between patients treated utilizing a linear accelerator versus a tri-60Co teletherapy platform.

OUTLINE:

Patients undergo SBRT every other day (QOD) for 14 days. Patients may also receive androgen deprivation therapy (ADT) comprised of a luteinizing hormone-releasing hormone agonist or a gonadotropin-releasing hormone antagonist, and an oral anti-androgen for 6 months at the discretion of the treating physician.

After completion of study treatment, patients are followed up at 1 month, every 3 months for 1 year, every 6 months for 4 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* History of histologically confirmed, clinical localized adenocarcinoma of the prostate treated with radical prostatectomy with definitive intent
* Presence of adverse pathologic features at the time of prostatectomy (positive surgical margin, pathologic T-stage 3-4 disease, pathologic Gleason score 8-10 disease, presence of tertiary Gleason grade 5 disease) OR documentation of rising prostate-specific antigen on at least two consecutive draws, with the magnitude of prostate-specific antigen exceeding 0.03 ng/mL
* Computed tomography (CT) scan and MRI of the pelvis within 120 days prior to enrollment (note: [a] if patient has medical contraindication to MRI, an exemption will be granted and enrollment can proceed [b] for patients with PSA < 1.0 ng/mL, the treatment planning CT can substitute for a diagnostic CT scan)
* Bone scan within 120 days prior to enrollment; if the bone scan is suspicious, a plain x-ray and/or MRI must be obtained to rule out metastasis, and advanced imaging (e.g., 18NaF positron emission tomography [PET]/CT) is strongly recommended
* Karnofsky performance score (KPS) >= 70
* Ability to understand, and willingness to sign, the written informed consent

Exclusion Criteria:

* Patients with any evidence of distant metastases
* Patients with pathologically-confirmed N1 prostate cancer
* Patients with neuroendocrine or small cell carcinoma of the prostate
* Prior cryosurgery, high-intensity focused ultrasound ablation (HIFU) or brachytherapy of the prostate
* Prior pelvic radiotherapy
* History of Crohn's disease, ulcerative colitis, or ataxia telangiectasia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Biochemical recurrence-free survival (BCRFS) | Up to 5 years
  Defined as serum prostate-specific antigen (PSA) rising from the post-treatment nadir to a level of 0.4 ng/mL or more with a confirmatory second test, initiation of salvage androgen deprivation therapy, or continued rise in PSA after stereotactic body radiation therapy (SBRT). The Kaplan-Meier product-limit estimate of the BCRFS will be estimated and presented graphically. One sample log-rank test will be used to test difference in BCRFS between intervention and historical control. The median BCRFS time will be calculated with 95% confidence interval. Summaries of the number and percentage of patients experiencing a biochemical recurrence will be provided.
Physician-scored toxicity | Up to 5 years
  Represented by the rates of acute (early, within 90 days of SBRT) and late (90 or more days after SBRT) genitourinary and gastrointestinal toxicity based on the Common Terminology Criteria for Adverse Events version 4.03. Adverse Events (AEs) and serious adverse events (SAEs) will be listed individually by patient.
Patient-reported toxicity outcomes EPIC-26 | Up to 5 years
  Patient-reported toxicity outcomes represented by changes in the urinary incontinence, urinary obstruction, bowel, sexual function, and hormone/vitality domains on the Expanded Prostate Cancer Index-26 (EPIC-26) quality of life instrument (scored from 0-100 points for each domain, higher scores reflect worse symptom/bother severity.)
Patient-reported toxicity outcomes IPSS | Up to 5 years
  Patient-reported toxicity outcomes represented by changes in International Prostate Symptom Scores (IPSS) (scored from 0-35 points, higher scores reflect worse symptom/bother severity.).

SECONDARY OUTCOMES:
Proportion of stereotactic body radiation therapy (SBRT) fractions for which on-line adaptive radiotherapy was utilized in the subset of patient treated with magnetic resonance imaging (MRI)-guided radiotherapy | Up to 5 years
  Point estimate and the corresponding 95% confidence interval will be calculated for the proportion of SBRT fractions for which on-line adaptive radiotherapy is required due to changes in organ-at-risk anatomy, in the subset of patients treated with MRI-guided radiotherapy.

OTHER OUTCOMES:
Physician-scored Toxicity profiles patients treated utilizing a linear accelerator | Up to 5 years
  Comparative analysis will be performed to assess physician-scored toxicity profiles for treated utilizing a linear accelerator. Unpaired t-test or Wilcoxon rank sum test will be used for quantitative toxicity metrics.
Patient-reported toxicity outcomes; patients treated utilizing a linear accelerator | Up to 5 years
  Comparative analysis will be performed to assess patient-reported toxicity profiles for treated utilizing a linear accelerator. Unpaired t-test or Wilcoxon rank sum test will be used for quantitative toxicity metrics.
Physician-scored toxicity profiles patients treated utilizing the magnetic resonance imaging (MRI)-guided device | Up to 5 years
  Comparative analysis will be performed to assess toxicity profiles with patients treated utilizing a linear accelerator. Chi-square test or Fisher's exact test will be used for qualitative toxicity measurements, while unpaired t-test or Wilcoxon rank sum test will be used for quantitative toxicity metrics.
Patient-reported toxicity profiles patients treated utilizing the magnetic resonance imaging (MRI)-guided device | Up to 5 years
  Comparative analysis will be performed to assess patient-reported toxicity profiles for treated utilizing an MRI-guided radiotherapy device. Unpaired t-test or Wilcoxon rank sum test will be used for quantitative toxicity metrics.

CONTACTS AND LOCATIONS:
Overall Officials: Amar Kishan, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (2):
- United States (2):
  - USC Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California

REFERENCES:
- [Derived] Nikitas J, Ballas LK, Romero T, Lynch C, Ma TM, Valle LF, Sachdeva A, Chong N, Basehart V, Franco A, Reiter R, Saigal C, Chamie K, Litwin MS, Donin NM, Rettig M, Nickols NG, Cao M, Liauw SL, Steinberg ML, Kishan AU. Patient-Reported Outcomes With Stereotactic Intensity Modulated Radiotherapy After Radical Prostatectomy: A Nonrandomized Clinical Trial. JAMA Oncol. 2025 Jul 1;11(7):726-734. doi: 10.1001/jamaoncol.2025.1059. PMID 40372727
- [Derived] Nikitas J, Smith LM, Gao Y, Ma TM, Sachdeva A, Yoon SM, Jiang T, Low DA, Ballas LK, Steinberg ML, Cao M, Kishan AU. The role of adaptive planning in margin-reduced, MRI-guided stereotactic body radiotherapy to the prostate bed following radical prostatectomy: Post-hoc analysis of a phase II clinical trial. Radiother Oncol. 2023 Jun;183:109631. doi: 10.1016/j.radonc.2023.109631. Epub 2023 Mar 18. PMID 36934894